CLINICAL TRIAL: NCT01720433
Title: Reduction of Pain Following Laparoscopic Surgery: A Double Blind Prospective Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northampton General Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Achal Khanna, Mr Achal Khanna Specialist Registrar - Surgery, Northampton General Hospital NHS Trust
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: lap pain trial NGH
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Post-operative Pain
Keywords: laparoscopic pain prospective blinded trial
MeSH Terms: conditions — Pain, Postoperative | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): In the intervention group, in addition to the above, the patient was placed in the Trendelenburg position (30°) and a pulmonary recruitment maneuver utilized, consisting of two manual inflations to a maximum pressure of 60 cm H2O. This was performed by the Anaesthetist, who held each positive pressure inflation for five seconds, with the valves on the operative ports fully open.
  Interventions: Procedure: intervention
- control arm (No Intervention): In the control group residual carbon dioxide pneumo-peritoneum was evacuated at the end of the procedure by passively allowing the abdomen to decompress by opening the operative ports.

INTERVENTIONS:
Procedure: intervention — The patient was placed in the Trendelenburg position (30°) and two manual lung inflations to a maximum pressure of 60 cm H2O for five seconds, with the valves on the operative ports fully open.
  Other Names: pulmonary recruitment maneouvre
  Arms: intervention

SUMMARY:
Shoulder tip and abdominal pain following laparoscopic procedures are well recognized as causes of post-operative morbidity. This prospective, double-blind, randomized controlled trial attempts to reduce post-operative pain in patients undergoing laparoscopic surgery by implementing a simple intra-operative technique.

Patients who undergo elective laparoscopic cholecystectomy for gallbladder disease or laparoscopic inguinal hernia repair will be recruited to the trial. Patients will be randomized to either the current standard (control group) or to receive an intervention to remove residual CO2. In the intervention group the pneumo-peritoneum will be removed, at the end of the operation, by placing the patient in the Trendelenburg position and utilising a pulmonary recruitment maneuver consisting of two manual inflations to a maximum pressure of 60 cm H2O. In the control group residual pneumo-peritoneum will be evacuated at the end of the procedure by passive decompression via the open operative ports.

DETAILED DESCRIPTION:
This trial recruited 76 randomly assigned patients, 37 in the intervention group and 39 in the control group. The overall post-surgery pain scores, as analysed by two-way ANOVA, were significantly lower in the intervention group (P=0.0019). On Bonferroni post-tests both 12 hour (P<0.01) and 24-hour (P<0.01) pain scores were significantly lower in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* All patients were recruited from a single Consultant's surgical clinic at the same District General Hospital between August 2010 and February 2012. This study was approved by the local ethics committee (National Research Ethics Service REC ref: 09/H0405/65) and informed consent was obtained from all patients after they had the opportunity to study information leaflets that were also given to them. The trial was designed as a prospectively randomized and double blind trial with a 1:1 (control:intervention) allocation.

The inclusion criteria was all adults with an American Society of Anesthesiologists (ASA) physical status grade 1 or 2, who were undergoing elective laparoscopic cholecystectomy for gallbladder disease or laparoscopic inguinal hernia repair performed as a transabdominal preperitoneal procedure (TAP). All procedures and data collection occurred at a District General Hospital.

Exclusion Criteria:

The pre-operative exclusion criteria included patients younger than 18 years, those who refused to give consent, those that had an inability to understand the research questionnaire and pregnancy. Patients who were found to require additional procedures, for example a conversion to open surgery, were excluded from the study prior to randomization.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
pain scores at varying time points pot operatively | 48 hours
  Pain scores were assessed by the use of a validated visual analogue score (whereby '0' was equivalent to 'no pain' and '10' equivalent to the worst 'conceivable pain.')

CONTACTS AND LOCATIONS:
Overall Officials: Achal Khanna, MRCSEd, Principal Investigator — Northampton General Hospital Northampton England
Locations (1):
- Northampton General Hopsital, Northampton, Northamptonshire, United Kingdom

REFERENCES:
- [Derived] Khanna A, Sezen E, Barlow A, Rayt H, Finch JG. Randomized clinical trial of a simple pulmonary recruitment manoeuvre to reduce pain after laparoscopy. Br J Surg. 2013 Sep;100(10):1290-4. doi: 10.1002/bjs.9202. PMID 23939841